CLINICAL TRIAL: NCT05967091
Title: Targeted Lung Denervation (TLD) With the Ryme Medical Lung Denervation System in Patients With Chronic Obstructive Pulmonary Disease (COPD) - Ryme Medical TLD Pilot Study
Brief Title: Ryme Medical TLD Pilot Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ryme Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-01
Record Dates: First submitted 2023-07-14; First posted 2023-08-01 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Dyspnea; Lung denervation; Bronchoscopic intervention; Lung disease; Lung diseases, obstructive; Respiratory tract diseases
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea; Lung Diseases; Lung Diseases, Obstructive; Respiratory Tract Diseases

STUDY DESIGN:
Intervention Model Description: Single-arm, non-randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Targeted Lung Denervation (Experimental): Targeted lung denervation (TLD) with the Ryme Medical Lung Denervation System
  Interventions: Device: Targeted Lung Denervation

INTERVENTIONS:
Device: Targeted Lung Denervation — Targeted Lung Denervation (TLD) is a bronchoscopically guided, minimally invasive procedure using the Ryme Medical Lung Denervation System
  Other Names: TLD

SUMMARY:
Targeted lung denervation (TLD) with the Ryme Medical Lung Denervation System in patients with chronic obstructive pulmonary disease (COPD) - Ryme Medical TLD Pilot Study

DETAILED DESCRIPTION:
The study is a prospective, multi-center, non-randomized study to evaluate the safety and performance of the Ryme Medical Lung Denervation System in patients with chronic obstructive pulmonary disease (COPD)

ELIGIBILITY:
Key Inclusion Criteria:

* Symptomatic chronic obstructive pulmonary disease
* ≥40 years of age
* Smoking history of at least 10 pack years
* Candidate for bronchoscopy in the opinion of the Investigator

Key Exclusion Criteria:

* Recent COPD exacerbation or respiratory infection
* Prior lung intervention with device in place
* Pulmonary nodule or malignancy requiring treatment
* Current chemotherapy or radiation therapy and/or has received treatment within 6 months
* Current smoker, using e-cigarettes or vaping, or taking any inhaled substances not prescribed by a physician
* Clinically significant serious or unstable medical conditions (e.g., heart disease requiring treatment, uncontrolled diabetes)
* Pregnant, nursing, or intent to become pregnant during study duration

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-06 (Actual); Primary Completion 2025-05-22 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Device Safety | 30 Days
  Serious adverse events associated with the Ryme Medical Lung Denervation System

SECONDARY OUTCOMES:
Device Success | Day 0
Technical Success | Day 0

CONTACTS AND LOCATIONS:
Locations (7):
- Australia (2):
  - Melbourne Health - The Royal Melbourne Hospital, Melbourne
  - Macquarie University, Sydney
- Karl Landsteiner Institute for Lung Research, Vienna, Austria
- Rigshospitalet, Copenhagen, Denmark
- Healthycore, Tbilisi, Georgia
- University of Groningen Medical Center, Groningen, Netherlands
- Royal Brompton, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No